CLINICAL TRIAL: NCT06777524
Title: Short-term and Long-term Effects of Skin-to-skin Contact in Healthy Term Infants
Brief Title: Skin-to-skin Contact in Healthy Term Infants
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Korea University Anam Hospital (Other)
Responsible Party: Principal Investigator, Juyoung Lee, Professor, Korea University Anam Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 2024AN0613
Record Dates: First submitted 2025-01-06; First posted 2025-01-16 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Skin-to-skin Contact
Keywords: skin-to-skin contact; infant; neurodevelopmental outcome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: * Randomization will be carried out by one investigator from the Department of Preventive Medicine, who does not have direct contact with the infants or their parents in the hospital.
  * A computer program will be used to randomly assign participants into two groups using permuted blocks (4 and 6), stratified by first-born and subsequent-born infants, with a 1:1 random allocation. The assigned groups will be communicated to the principal investigator.
  * Parents will not be informed of their assigned group, and the study will be described as an investigation on the infant's sleep, feeding, bonding, and overall health, so as not to influence the mother-infant contact time.
  * All personnel responsible for scoring and evaluating the outcomes will also be blinded to group allocation, except for the researchers who provide education to the control and intervention groups. To ensure proper allocation concealment, the randomization sequence will remain concealed until the study is completed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- control group (No Intervention): Parents of the control group will receive general education about sleep, breastfeeding, and bathing, which are provided to parents before going home after birth.
- skin-to-skin contact (SSC) group (Experimental): For the intervention group, additional education on the importance and clinical benefits of mother-infant skin-to-skin contact will be provided (including an educational video).
  Interventions: Behavioral: skin-to-skin contact education

INTERVENTIONS:
Behavioral: skin-to-skin contact education — For the intervention group, additional education on the importance and clinical benefits of mother-infant skin-to-skin contact will be provided (including an educational video). They will be instructed to engage in a minimum of 6 hours of skin-to-skin contact per day with the infant's and mother's chests exposed for at least 15 minutes per session, and to keep a record of the contact time, as well as the time spent holding the clothed infant and a daily feeding diary.
  Arms: skin-to-skin contact (SSC) group

SUMMARY:
This is a prospective, double-blind, randomized controlled clinical trial study to investigate short- and long-term effects of mother-infant skin-to-skin contact in healthy term infants, in order to provide supporting data for emphasizing mother-infant skin contact and family-centered care in South Korea.

ELIGIBILITY:
Inclusion Criteria:

* Babies born at Korea University Anam Hospital
* Term infants (37 weeks or more)
* Infants with a birth weight of 2,500g or more
* Healthy infants with an Apgar score of 7 or higher at 5 minutes
* Mothers and infants without severe acute complications, such as requiring intensive care treatment immediately after delivery

Exclusion Criteria:

* Preterm infants born at 37 weeks of less gestation
* Low birth weight infants weighing less than 2500g at birth
* Mothers under the age of 20
* Unmarried mothers
* Multiple pregnancies (twins or triplets)
* Parents do not consent to participation in the study

Ages: 1 Hour to 72 Hours | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 130 (Estimated)
Dates: Start 2025-02-10 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2030-01-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of any breast feeding (combined with formula and/or solid or not) | at 4 months of age
  This includes both exclusive breastfeeding and partial breastfeeding combined with formula and/or solid food.

SECONDARY OUTCOMES:
Percentage of any breast feeding (combined with formula and/or solid or not) | at 1 month, 8 months, and 12 months of age
  This includes both exclusive breastfeeding and partial breastfeeding combined with formula and/or solid food.
Korean-Edinburgh Postnatal Depression score | 3 to 7 days, 1 month, and 4 months of infant age
  mother questionnaire range 0-30 low risk 0-8 borderline risk 9-12 high risk 13-30
Parent State-Trait Anxiety Inventory score | 3 to 7 days, 1 month, 4 months, 8 months, and 12 months of infant age
  mother questionnaire range 20-80 no or low anxiety 20-37 moderate anxiety 38-44 high anxiety 45-80
Maternal Postnatal Attachment Scale score | at 1 month, 4 months, 8 months, and 12 months of infant age
  mother questionnaire The score in the questionnaire ranges from 19 to 95, with a higher score indicating greater parent-infant attachment.
Artificial intelligence (AI) analysis for infant general movement videos | at 3-6 days, 1 and 4 months of age
  AI algorithms will be developed for analyzing infant movement captured in video. For this, computer vision techniques will be used for tracking joint movement and extracting relevant features. Machine learning models will then be trained to identify deviation from typical movement patterns, and system's performance will be evaluated using long-term development outcome measures.
Developmental Screening (K-DST) score | at 4, 8, 12, 24 and 36 months of infant age
  mother questionnaire, score of each developmental area K-DST has 6 domains; gross motor, fine motor, cognition, language, social skills, and self-help.
  The total score was evaluated based on the transfer points of each domain. The K- DST results are broadly grouped into 5 categories: (1) good, (2) requires follow-up examination, (3) requires detailed assessment, (4) continued care, and (5) other.
Infant temperament measured by Korean-Infant Behavior Questionnaire-Revised (K-IBQ-R) | at 8 months
  IBQ assessed 6 domains of infant temperament (activity level, soothability, fear, distress to limitations, smiling and laughter, and duration of orienting).The items on the IBQ ask parents to rate the frequency of specific temperament-related behaviors observed over the past week.
Korean-Early Childhood Behavior Questionnaire-Revised (K-ECBQ-R) | at 24months
  The Early Childhood Behavior Questionnaire (ECBQ) is a parent-report tool used to assess temperament in young children, based on observable behaviors. It includes 201 items grouped into 18 fine-grained subscales, which are further organized into three broad temperament factors
  1. Surgency - Reflects high energy and positive emotions (e.g., impulsivity, activity level, high-intensity pleasure, sociability and positive anticipation)
  2. Negative Emotionality - Captures sensitivity to negative experiences (e.g., discomfort, fear, motor activation, sadness, perceptual sensitivity, shyness, soothability and frustration scales).
  3. Effortful Control - Represents self-regulation and attention skills (e.g.,inhibitory control, attention shifting, low-intensity pleasure, cuddliness and attention focusing).
Bayley Scales of Infant Development III | at 24 months, and 36 months of infant age
  scale scores for each development areas (cognitive, language, motor) score range : 0-200 above average (1-2 SD, score 116-130) average ( 1 to 1 SD, score 85-115) below average (1 to-2 SD, score 84-70) well below average (<-2 SD, scores < 70).
Sequenced Language Scale for Infant (SELSI) | at 24 months, and 36 months of infant age
  percentile of each area (receptive and expressive language abilities). the raw scores is classified in accordance with standard guidelines: average, within -1 SD of the mean; mild delay, up to -2 SD; and delay, >-2 SDs below the mean scores.
Modified Checklist for Autism in Toddlers (M-CHAT) | at 24 months, and 36 months of infant age
  mother questionnaire total score 0-2: low risk total score 3-7: moderate risk total score 8-20: high risk
Child Behavior Checklist (CBCL) | at 24 and 36 months of age
  behavior screening questionnaire result t-score ≤ 59: non-clinical symptoms, t-score between 60 and 64: at risk for problem behaviors t-score ≥ 65: clinical symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- Korea University Anam Hospital NICU, Seoul, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Yes
Collected data will be available upon request from the corresponding author after completion of the study.
Supporting Information: Study Protocol, SAP, ICF, CSR

REFERENCES:
- [Derived] Cho H, Park J, Choe SA, Lee J. Short-term and long-term effects of skin-to-skin contact in healthy term infants: study protocol for a parallel-group double-blind randomised controlled trial. BMJ Open. 2025 Oct 14;15(10):e104809. doi: 10.1136/bmjopen-2025-104809. PMID 41087107